CLINICAL TRIAL: NCT04495959
Title: Dynamic Whole Body Positron Emission Tomography/ Magnetic Resonance Imaging
Brief Title: Dynamic Whole Body PET/ MRI
Status: Withdrawn | Type: Observational
Why Stopped: Study never initiated, should have been removed prior to last update.
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Sponsor
Other Study IDs: H20-02418
Record Dates: First submitted 2020-07-24; First posted 2020-08-03 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-11

CONDITIONS: Prostatic Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- 68Ga-HTK03149 PET/MRI DWB scan: All participants will undergo the same procedures listed in "Detailed Description" in the protocol section.
  Interventions: Drug: 68Ga-HTK03149

INTERVENTIONS:
Drug: 68Ga-HTK03149 — PET/MRI scan with radiotracer 68Ga-HTK03149

SUMMARY:
Prostate cancer is the third most common cause of cancer death in men. Most patients with localized prostate cancer will be cured with surgery or radiation therapy, but up to 35% of patients will have their prostate cancer return.Current conventional imaging modalities have limitations particularly at low prostate specific antigen levels. This study proposes to use 68Ga-HTK03149 Dynamic Whole Body (DWB) Positron Emission Tomography / Magnetic Resonance Imaging (PET/MRI) scans which targets prostate-specific membrane antigens (PSMA) to detect where in the body the prostate cancer has recurred.

DETAILED DESCRIPTION:
This is a prospective registry study to evaluate the diagnostic utility of 68Ga-HTK03149 DWB PET/MRI to stage patients with high risk prostate cancer who will subsequently under go radical prostatectomy.

Eligible subjects will undergo a 68Ga-HTK03149 DWB PET/MRI at the University of British Columbia (UBC) - Vancouver, Djavad Mowafaghian Centre for Brain Health where the UBC PET/MRI is located. Each subject will receive a 18F-DCFPyL PET/MRI DWB scan at the UBC centre, as part of this research study. Each study subject will receive a bolus intravenous dose of 18F-DCFPyL. The subject will be placed on the PET/MRI scanner for a dynamic whole body PET scan. Then after a brief break off the scanner, they will return to the scanner for the standard whole body PET/MRI scan.

The PET/MRI scan will take approximately 3.5 hours of patient time above and beyond the time needed for standard of care.

Medical History Questionnaire: Demographic and medical history data will be collected either in person before the PET scan appointment or by mail or phone, whichever is the most convenient to the subject.

Follow-up assessments: All subjects will be contacted by phone the day after the injection of 68Ga-HTK03149. The subjects will be asked if they experienced any undesirable effects during the 12 hours after the administration of 68Ga-HTK03149. The local site attending nuclear medicine physician will then make an assessment as to whether these effects are likely related to 68Ga-HTK03149 administration.

All subjects will be followed for 5 years following the 68Ga-HTK03149 PET/CT exam to assess the presence of recurrence. The evaluation will include a chart review of available imaging, laboratory tests, and treatment. The data required can be obtained from a review of the patient's paper and electronic charts, supplemented by telephone contact as needed to complete the information.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with biopsy-proven high risk prostate cancer (UCSF/CAPRA score 6 or higher) scheduled for radical prostatectomy.
* Able to not use the washroom for the duration of the dynamic imaging scanning.
* Eastern Cooperative Oncology Group performance status of 2 or less.
* Able to lie supine for the required duration of the scans

Exclusion Criteria:

* Meet the exclusion criteria for the appropriate standard of care imaging.
* Experience claustrophobia.
* Subjects with severe renal disease or acutely deteriorating renal function (eGRF<30 mL/min)
* Subjects may not take part in this study if they have a pacemaker, an implanted defibrillator, or certain other implanted electronic or metallic devices, shrapnel, or other metal.

Ages: 19 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed high risk prostate cancer (UCSF/CAPRA score of 6 or higher) who are scheduled to undergo radical prostatectomy.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of Dynamic Whole Body 68Ga-HTK03149PET/MRI imaging in the assessment of high risk prostate cancer. | 5 years after 68Ga-HTK03149DWB PET/MRI scan
  Determination of sensitivity when compared with pathology reports

SECONDARY OUTCOMES:
Accuracy of combined DWB PET/MRI to assess the extent of prostate cancer | 5 years after 68Ga-HTK03149 DWB PET/MRI scan
  Comparison of parametric images derived from dynamic whole body PET imaging to conventional static PET images as well as MRI images . Assessment as to whether parametric images are able to distinguish normal organ accumulation (e.g. ureters, kidneys, bladder, bowel) from tumour uptake, based on the kinetics of radiotracer accumulation. Quantitative comparison of image contrast and signal-to-noise ratio (SNR) between static and parametric images from dynamic scans will be completed.
Number of participants with self-reported 68Ga-HTK03149 related adverse event | 12 hours post 68Ga-HTK03149 injection
  Patients will be contacted by phone the day after the 68Ga-HTK03149PET/CT scan to see if they experienced any adverse events in the 12 hours following the 18F-DCFPyL injection. These are recorded and evaluated for severity and likelihood they are related to the study drug. All adverse events will be recorded and summarized in the final report.

CONTACTS AND LOCATIONS:
Locations (1):
- BC Cancer, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
no plan